CLINICAL TRIAL: NCT04147442
Title: A Clinical Investigation Comparing a Standard Hearing Aid Fitting Protocol and a Fitting Protocol Optimized for Musicians
Brief Title: A Standard Music Program Compared to an Optimized Music Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bernafon AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BF006-1902
Record Dates: First submitted 2019-10-09; First posted 2019-11-01 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: The participants will have access to both music programs for 10 +/- 7 days. During this time they will use both programs and switch between them during music playing situations.
Masking Description: The allotted program position for the music programs will be randomized. Half of the participants will have the fine-tuned program in slot 2 and half will have it in slot 3. They will not know in which position the fine-tuned program is versus the standard program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music program fine-tuned and standard (Experimental): The fine-tuned program and the standard program will be compared within the same instrument as a hearing aid can have up to 4 different listening programs in it.
  Interventions: Device: Hearing aid with fine-tuned and standard programs

INTERVENTIONS:
Device: Hearing aid with fine-tuned and standard programs — A digital, wireless hearing aid is programmed specifically to each subject's hearing loss and fitted with both a program that is fine-tuned for their specific music playing as well as the standard music program that uses pre-determined settings.
  Other Names: Viron 9 mini receiver-in-the-ear hearing aid

SUMMARY:
The trial will test whether a standard music program that is an offset to the general program provides the same benefit as a music program that is individually customized for each test participant. The trial seeks to investigate the benefit received by musicians that regularly play an instrument and belong to an organized music group or orchestra instead of people that listen to music.

DETAILED DESCRIPTION:
The initial goal of hearing aids is to amplify speech and facilitate speech understanding especially in noise. Besides speech difficulty, people with hearing loss also report a reduced enjoyment of music. The hearing aid settings used for amplifying speech often have adverse effects on music.

For this study, the sponsor will carry out testing with participants with hearing loss to compare dedicated music programs. The current study will compare the standard music program available in the software to one that is fine-tuned for each subject. The hearing aids that will be used for the study are certified by the European Conformity and have been on the market for almost one year. The goal is to determine whether musicians will perceive a difference and prefer a fine-tuned music program over the default music program in real-life situations.

ELIGIBILITY:
Inclusion Criteria:

* All classifications of hearing loss (sensorineural, conductive, mixed)
* If conductive or mixed, approval for amplification by a physician is needed
* All shapes of hearing loss (flat, sloping, reverse slope, notch)
* Severity ranging from mild to profound
* German or French speaking
* Play a musical instrument
* Ability and willingness to sign the consent form

Exclusion Criteria:

* Normal hearing
* Contraindications for amplification
* Active ear disease
* Don't play an instrument
* Inability to follow the study procedures due to language problems, psychological disorders, dementia, or other cognitive problems
* Unable to attend study appointments due to reduced mobility
* Reduced ability to describe auditory impressions and usage of hearing aids
* Uncooperative so that it is ot possible to record a valid audiogram
* Severely reduced dexterity
* Central hearing disorders
* Sponsor employees
* Family members of employees of the Sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Simon, AuD, Principal Investigator — Bernafon AG
Locations (1):
- Bernafon AG, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Music Program Fine-tuned and Standard: The fine-tuned program and the standard program will be compared within the same instrument as a hearing aid can have up to 4 different listening programs in it.
  The hearing aid is a digital, wireless hearing aid that is programmed specifically to each subject's hearing loss and fitted with two programs. One is fine-tuned for their specific music playing and one is the standard music program based on pre-determined settings.
Period: Overall Study
Arm/Group | Music Program Fine-tuned and Standard
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Music Program Fine-tuned: The fine-tuned program and the standard program will be compared within the same instrument as a hearing aid can have up to 4 different listening programs in it.
  Hearing aid with fine-tuned program: A digital, wireless hearing aid that is programmed specifically to each subject's hearing loss and fine-tuned for their specific music playing.
Arm/Group | Music Program Fine-tuned
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 67 [24 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 20
Hearing Loss [Mean (Standard Deviation); unit: decibels] | 46 (16)

OUTCOME MEASURES:

1. Primary Outcome: Preference Rating
Description: Subjects will answer a questionnaire that asks them to choose which program that they preferred. The questionnaire gives Program 1 or Program 2 as the choices as well as a no Preference option for those that did not notice a difference between the two. The percentage of subjects that chose each Program will be calculated to determine if more preferred the optimized music program.
Time Frame: 20 days
Population: There were 15 males and 5 females ranging in age from 24 to 81 years with a mean age of 67. The mean average Hearing loss was 46 dB HL with a standard deviation of 16 dB HL.
Measure: Count of Participants; unit: Participants
Arm/Group | Music Program Fine-tuned and Standard
Number analyzed (Participants) | 20
Participants
  Fine-tuned Preference | 14
  Standard Preference | 3
  No Preference | 3

2. Secondary Outcome: Sound Perception Test - Pitch
Description: The sound perception test is called the Adaptive Music Perception test. It is tested in the lab with digitally synthesized recordings of components of tones. It tests the overall perception of Meter with pitch (in Hz). A lower score is better. A higher score means that it took higher Levels of Hz to perceive a difference between musical notes.The subjects are tested in the unaided, aided with the standard program, and aided with the test (optimized) program. The scores will be averaged and analyzed to determine if one program results in better (lower) test scores.
Time Frame: 0,10, and 20 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hertz
Groups:
- Music Program Fine-tuned: The hearing aid is a digital, wireless hearing aid that is programmed specifically to each subject's hearing loss and fitted with two programs. One is fine-tuned for their specific music playing and one is the standard music program based on pre-determined settings.
  They will perform the test with the fine-tuned program.
- Music Standard Program: The hearing aid is a digital, wireless hearing aid that is programmed specifically to each subject's hearing loss and fitted with two programs. One is fine-tuned for their specific music playing and one is the standard music program based on pre-determined settings.
  They will perform the test with the standard default music program.
- Unaided: The participants will perform the test with no hearing aids.
Arm/Group | Music Program Fine-tuned | Music Standard Program | Unaided
Number analyzed (Participants) | 20 | 20 | 20
hertz | 1.4 (0.7) | 1.8 (0.6) | 1.9 (0.8)

3. Secondary Outcome: Music Sound Quality Rating
Description: The sound quality of the devices when listening/playing music will be rated using a questionnaire. The questionnaire asks subjects to rate various aspects of the sound using a 5-point scale with 1 being the worst answer and 5 being the best. The questionnaire will be answered for Program 1 and Program 2. The scores for each question will be averaged across subjects and the difference between the two programs calculated to determine if one music program results in better sound quality scores. A positive score is in favor of the fine-tuned program and a negative score would be in favor of the standard program. They will test Program 1 and Program 2 during the same period as they have the ability to use a button on the Hearing aid to switch between programs.
Time Frame: 0,10, and 20 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Music Program Fine-tuned and Standard
Number analyzed (Participants) | 20
units on a scale
  Sound Quality-pleasant | 0.66 (0.37)
  Sound Quality-natural | 0.69 (0.35)

4. Other Pre Specified Outcome: Occurrence of Device Related Adverse Events
Description: The number of Device Related Adverse Events will be monitored and totaled. Each Adverse Event is measured using a severity scale of: mild, moderate, or severe. The causality is measured with a scale of: Not related, unlikely, possible, probable, and causal relationship.
Time Frame: 0,10, and 20 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Music Program Fine-tuned and Standard
Number analyzed (Participants) | 20
Participants | 0

5. Secondary Outcome: Sound Perception Test - Duration
Description: The sound perception test is called the Adaptive Music Perception test. It is tested in the lab with digitally synthesized recordings of components of tones. It tests the overall perception of duration (in milliseconds). A lower score is better. A higher score means that it took longer in milliseconds to perceive a difference between musical notes.The subjects are tested in the unaided, aided with the standard program, and aided with the test (optimized) program. The scores will be averaged and analyzed to determine if one program results in better (lower) test scores.
Time Frame: 0,10, and 20 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Music Program Fine-tuned: The hearing aid is a digital, wireless hearing aid that is programmed specifically to each subject's hearing loss and fitted with two programs. One is fine-tuned for their specific music playing and one is the standard music program based on pre-determined settings.
  The participants will perform the test with the fine-tuned music program.
- Music Standard Program: The hearing aid is a digital, wireless hearing aid that is programmed specifically to each subject's hearing loss and fitted with two programs. One is fine-tuned for their specific music playing and one is the standard music program based on pre-determined settings.
  The participants will perform the test with the standard default music program.
Arm/Group | Music Program Fine-tuned | Music Standard Program | Unaided
Number analyzed (Participants) | 20 | 20 | 20
milliseconds | 31 (22) | 39 (24) | 35 (21)

6. Secondary Outcome: Sound Perception Test - Level
Description: The sound perception test is called the Adaptive Music Perception test. It is tested in the lab with digitally synthesized recordings of components of tones. It tests the overall perception of Meter with Level (in decibels). A lower score is better. A higher score means that it took higher levels in dB to perceive a difference between musical notes.The subjects are tested in the unaided, aided with the standard program, and aided with the test (optimized) program. The scores will be averaged and analyzed to determine if one program results in better (lower) test scores.
Time Frame: 0,10, and 20 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: decibels
Groups:
- Music Program Fine-tuned: The hearing aid is a digital, wireless hearing aid that is programmed specifically to each subject's hearing loss and fitted with two programs. One is fine-tuned for their specific music playing and one is the standard music program based on pre-determined settings.
  The participants performed the test with the fine-tuned music program.
- Music Program Standard: The hearing aid is a digital, wireless hearing aid that is programmed specifically to each subject's hearing loss and fitted with two programs. One is fine-tuned for their specific music playing and one is the standard music program based on pre-determined settings.
  The participants performed the test with the standard default music program.
- Unaided: The participants performed the test with no hearing aids.
Arm/Group | Music Program Fine-tuned | Music Program Standard | Unaided
Number analyzed (Participants) | 20 | 20 | 20
decibels | 1.5 (0.7) | 1.7 (0.5) | 1.9 (1.0)

7. Secondary Outcome: Sound Perception Test - Brightness
Description: The sound perception test is called the Adaptive Music Perception test. It is tested in the lab with digitally synthesized recordings of components of tones. The perception of the Timber of music is tested by the brightness (measured in dB). Lower scores are better. A higher score means that it took higher levels in dB to perceive a difference between musical notes.The subjects are tested in the unaided, aided with the standard program, and aided with the test (optimized) program. The scores will be averaged and analyzed to determine if one program results in better (lower) test scores.
Time Frame: 0,10, and 20 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | Music Program Fine-tuned | Music Program Standard | Unaided
Number analyzed (Participants) | 20 | 20 | 20
decibels | 0.4 (0.2) | 0.3 (0.2) | 0.5 (0.2)

8. Secondary Outcome: Sound Perception Test - Attack
Description: The sound perception test is called the Adaptive Music Perception test. It is tested in the lab with digitally synthesized recordings of components of tones. The perception of the Timber of music is tested by the attack (measured in Hz). Lower scores are better. A higher score means that it took higher levels in Hz to perceive a difference between musical notes.The subjects are tested in the unaided, aided with the standard program, and aided with the test (optimized) program. The scores will be averaged and analyzed to determine if one program results in better (lower) test scores.
Time Frame: 0,10, and 20 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hertz
Arm/Group | Music Program Fine-tuned | Music Program Standard | Unaided
Number analyzed (Participants) | 20 | 20 | 20
hertz | 158 (78.8) | 207.8 (97.8) | 197 (66.3)

9. Secondary Outcome: Sound Perception Test - Spectral Irregularities
Description: The sound perception test is called the Adaptive Music Perception test. It is tested in the lab with digitally synthesized recordings of components of tones. The perception of the Timber of music is tested by the spectral irregularities (measured in dB). Lower scores are better. A higher score means that it took higher levels in dB to perceive a difference between musical notes.The subjects are tested in the unaided, aided with the standard program, and aided with the test (optimized) program. The scores will be averaged and analyzed to determine if one program results in better (lower) test scores.
Time Frame: 0,10, and 20 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | Music Program Fine-tuned | Music Program Standard | Unaided
Number analyzed (Participants) | 20 | 20 | 20
decibels | 5 (2) | 4 (2) | 5 (2)

ADVERSE EVENTS:
Time Frame: 1 month
Description: Definition of adverse Events does not differ. Subjects are questioned at each Appointment to determine whether an adverse Event occurred outside of the clinic during the field trials.
Arm/Group | Music Program Fine-tuned
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Music Program Fine-tuned (N=20)
Cold (Infections and infestations) | 1 (20) — Subject had a common cold with nasal congestion and sneezing. No Fever or coughing was reported.
Foot Injury (Injury, poisoning and procedural complications) | 1 (20) — Subject injured foot while Walking. It healed by itself and did not require any Treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT04147442/Prot_001.pdf
  • Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT04147442/SAP_000.pdf